CLINICAL TRIAL: NCT01729208
Title: A Multicentre Dispensing Clinical Evaluation of MiSight® Lenses
Brief Title: An Evaluation of the Effectiveness of Dual Focus Soft Contact Lenses in Slowing Mypoia Progression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Collaborators: Visioncare Research Ltd. (Other)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CVI08008
Record Dates: First submitted 2012-11-14; First posted 2012-11-20 (Estimated); Results first posted 2020-02-24 (Actual); Last update posted 2020-02-24 (Actual); Status verified 2020-02

CONDITIONS: Myopia
Keywords: myopia progression; myopia control
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Dual Focus Soft Contact Lens (Experimental): Dual Focus Soft Contact Lens
  Interventions: Device: Dual Focus Soft Contact Lens
- Single Vision Soft Contact Lens (Placebo Comparator): Single Vision Soft Contact Lens
  Interventions: Device: Single Vision Soft Contact Lens

INTERVENTIONS:
Device: Dual Focus Soft Contact Lens
  Arms: Dual Focus Soft Contact Lens
Device: Single Vision Soft Contact Lens
  Arms: Single Vision Soft Contact Lens

SUMMARY:
The purpose of this study is to determine whether a new type of soft contact lens with a unique optical design (dual focus) is effective at slowing the progression of myopia (near-sightedness) in children.

DETAILED DESCRIPTION:
Subjects were randomized to wear test or control soft contact lens to determine whether a new type of soft contact lens with a unique optical design (dual focus) is effective at slowing the progression of myopia (near-sightedness) in children.

ELIGIBILITY:
Inclusion Criteria:

* Be between 8 and 12 years of age inclusive.
* Best-corrected visual acuity by manifest refraction of +0.10 logMAR.
* Spherical Equivalent Refractive Error between -0.75 and -4.00 D
* inclusive astigmatism: < -0.75 D and anisometropia: < 1.00 D
* Possess wearable and visually functional eyeglasses.
* Agree to wear the assigned contact lenses for a minimum of 10 hours per day, - at least 6 days per week, for the duration of the 3 year study.

Exclusion Criteria:

* Subject has previously or currently wears contact lenses or rigid gas permeable contact lenses, including orthokeratology lenses.
* Subject is currently or within 30 days prior to this study has been an active participant in another clinical study.
* Current or prior use of bifocals, progressive addition lenses, atropine, pirenzepine or ANY other myopia control treatment.
* Regular use of ocular medications (prescription or over-the-counter), artificial tears, or wetting agents.
* Current use of systemic medications which may significantly affect contact lens wear, tear film production, pupil size, accommodation or refractive state.
* A known allergy to fluorescein, benoxinate, proparacaine or tropicamide.
* Strabismus by cover test at far (4 m) or near (40 cm) wearing distance correction.
* Any ocular, systemic or neuro-developmental conditions that could influence refractive development.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 144 (Actual)
Dates: Start 2012-11 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2019-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: José Manuel González-Méijome, Principal Investigator — University of Minho
Locations (4):
- University of Waterloo School of Optometry, Waterloo, Ontario, Canada
- University of Minho Clinical & Experiment Optometry Research Lab, Braga, Portugal
- National University of Singapore Faculty of Medicine, Singapore, Singapore
- Aston University Ophthalmic Research Group, Birmingham, United Kingdom

REFERENCES:
- [Derived] Chamberlain P, Hammond DS, Bradley A, Arumugam B, Richdale K, McNally J, Hunt C, Young G. Eye growth and myopia progression following cessation of myopia control therapy with a dual-focus soft contact lens. Optom Vis Sci. 2025 May 1;102(5):353-358. doi: 10.1097/OPX.0000000000002244. Epub 2025 Mar 24. PMID 40132119
- [Derived] Chamberlain P, Bradley A, Arumugam B, Hammond D, McNally J, Logan NS, Jones D, Ngo C, Peixoto-de-Matos SC, Hunt C, Young G. Long-term Effect of Dual-focus Contact Lenses on Myopia Progression in Children: A 6-year Multicenter Clinical Trial. Optom Vis Sci. 2022 Mar 1;99(3):204-212. doi: 10.1097/OPX.0000000000001873. PMID 35086120
- [Derived] Chamberlain P, Peixoto-de-Matos SC, Logan NS, Ngo C, Jones D, Young G. A 3-year Randomized Clinical Trial of MiSight Lenses for Myopia Control. Optom Vis Sci. 2019 Aug;96(8):556-567. doi: 10.1097/OPX.0000000000001410. PMID 31343513

RESULTS

PARTICIPANT FLOW:
Period: Baseline
Arm/Group | Dual Focus Soft Contact Lens | Single Vision Soft Contact Lens
Started | 70 | 74
Completed | 65 | 70
Not Completed | 5 | 4
Not completed — Physician Decision | 5 | 4
Period: 12 Months Follow-up
Arm/Group | Dual Focus Soft Contact Lens | Single Vision Soft Contact Lens
Started | 65 | 70
Completed | 58 | 60
Not Completed | 7 | 10
Not completed — Withdrawal by Subject | 4 | 7
Not completed — Lost to Follow-up | 3 | 3
Period: 24 Months Follow-up
Arm/Group | Dual Focus Soft Contact Lens | Single Vision Soft Contact Lens
Started | 58 | 60
Completed | 55 | 60
Not Completed | 3 | 0
Not completed — Lost to Follow-up | 3 | 0
Period: 36 Months Follow-up
Arm/Group | Dual Focus Soft Contact Lens | Single Vision Soft Contact Lens
Started | 55 | 60
Completed | 52 | 56
Not Completed | 3 | 4
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 2 | 4

BASELINE CHARACTERISTICS:
Population: Subjects were randomized to wear dual focus soft contact lens and single vision soft contact lens.
Groups:
- Total: Total of all reporting groups
Arm/Group | Dual Focus Soft Contact Lens | Single Vision Soft Contact Lens | Total
Number analyzed (Participants) | 70 | 74 | 144
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 70 | 74 | 144
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.1 (1.3) | 10.1 (1.4) | 10.1 (1.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 37 | 69
  Male | 38 | 37 | 75
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 39 | 40 | 79
  East Asian | 16 | 18 | 34
  Indian/Pakistani/Sri Lankan | 5 | 7 | 12
  Other | 2 | 4 | 6
  Mixed | 8 | 5 | 13
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 32 | 32 | 64
  Singapore | 15 | 16 | 31
  United Kingdom | 13 | 15 | 28
  Portugal | 10 | 11 | 21

OUTCOME MEASURES:

1. Primary Outcome: Change in Refractive Error Relative to Baseline
Description: Mean change in refractive error, measured with cycloplegic auto-refraction in Diopters at 12 months, relative to baseline.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: Diopters
Units Other Than Participants: Eyes
Arm/Group | Dual Focus Soft Contact Lens | Single Vision Soft Contact Lens
Number analyzed (Participants) | 58 | 60
Number analyzed (Eyes) | 116 | 120
Diopters | -0.18 (0.39) | -0.58 (0.41)

2. Primary Outcome: Change in Refractive Error Relative to Baseline
Description: Mean change in refractive error, measured with cycloplegic auto-refraction in Diopters at 24 months, relative to baseline.
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: Diopters
Units Other Than Participants: Eyes
Arm/Group | Dual Focus Soft Contact Lens | Single Vision Soft Contact Lens
Number analyzed (Participants) | 55 | 60
Number analyzed (Eyes) | 110 | 120
Diopters | -0.38 (0.52) | -0.92 (0.53)

3. Primary Outcome: Change in Refractive Error Relative to Baseline
Description: Mean change in refractive error, measured with cycloplegic auto-refraction in Diopters at 36 months, relative to baseline.
Time Frame: 36 months
Measure: Mean (Standard Deviation); unit: Diopters
Units Other Than Participants: Eyes
Arm/Group | Dual Focus Soft Contact Lens | Single Vision Soft Contact Lens
Number analyzed (Participants) | 52 | 56
Number analyzed (Eyes) | 104 | 112
Diopters | -0.51 (0.64) | -1.24 (0.61)

4. Primary Outcome: Change in Axial Length Relative to Baseline
Description: Mean change in axial length measurement, in millimeters at 12 months, relative to baseline.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: Eyes
Arm/Group | Dual Focus Soft Contact Lens | Single Vision Soft Contact Lens
Number analyzed (Participants) | 58 | 60
Number analyzed (Eyes) | 116 | 120
mm | 0.09 (0.13) | 0.24 (0.15)

5. Primary Outcome: Change in Axial Length Relative to Baseline
Description: Mean change in axial length measurement, in millimeters at 24 months, relative to baseline.
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: Eyes
Arm/Group | Dual Focus Soft Contact Lens | Single Vision Soft Contact Lens
Number analyzed (Participants) | 55 | 60
Number analyzed (Eyes) | 110 | 120
mm | 0.21 (0.22) | 0.45 (0.23)

6. Primary Outcome: Change in Axial Length Relative to Baseline
Description: Mean change in axial length measurement, in millimeters at 36 months, relative to baseline.
Time Frame: 36 months
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: Eyes
Arm/Group | Dual Focus Soft Contact Lens | Single Vision Soft Contact Lens
Number analyzed (Participants) | 52 | 56
Number analyzed (Eyes) | 104 | 112
mm | 0.30 (0.28) | 0.62 (0.30)

7. Secondary Outcome: Number of Participants With Biomicroscopic Findings Greater Than Grade 2
Description: Cumulative incidence of biomicroscopic findings. Slit lamp severity greater than Grade 2 (based on a 0-4 scale, where 0=none and 4=severe).
Time Frame: Baseline
Measure: Number; unit: participants
Arm/Group | Dual Focus Soft Contact Lens | Single Vision Soft Contact Lens
Number analyzed (Participants) | 70 | 74
participants
  Corneal Staining | 0 | 0
  Conjuctival Staining | 0 | 0
  Bulbar Hyperemia | 0 | 0
  Limbal Hyperemia | 0 | 0
  Palpebral Hyperemia | 0 | 0
  Palpebral Roughness | 0 | 0
  Vascularization | 0 | 0
  "Other" Findings | 0 | 0

8. Secondary Outcome: Number of Participants With Biomicroscopic Findings Greater Than Grade 2
Description: as for outcome 7
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | Dual Focus Soft Contact Lens | Single Vision Soft Contact Lens
Number analyzed (Participants) | 58 | 60
participants
  Corneal Staining | 0 | 0
  Conjuctival Staining | 0 | 0
  Bulbar Hyperemia | 0 | 0
  Limbal Hyperemia | 0 | 0
  Palpebral Hyperemia | 0 | 0
  Palpebral Roughness | 1 | 0
  Vascularization | 0 | 0
  "Other" Findings | 0 | 0

9. Secondary Outcome: Number of Participants With Biomicroscopic Findings
Description: as for outcome 7
Time Frame: 24 months
Measure: Number; unit: participants
Arm/Group | Dual Focus Soft Contact Lens | Single Vision Soft Contact Lens
Number analyzed (Participants) | 55 | 60
participants
  Corneal Staining | 0 | 0
  Conjuctival Staining | 0 | 0
  Bulbar Hyperemia | 0 | 0
  Limbal Hyperemia | 0 | 0
  Palpebral Hyperemia | 0 | 0
  Palpebral Roughness | 0 | 0
  Vascularization | 0 | 0
  "Other" Findings | 0 | 0

10. Secondary Outcome: Number of Participants With Biomicroscopic Findings Greater Than Grade 2.
Description: as for outcome 7
Time Frame: 36 months
Measure: Number; unit: participants
Arm/Group | Dual Focus Soft Contact Lens | Single Vision Soft Contact Lens
Number analyzed (Participants) | 52 | 56
participants
  Corneal Staining | 0 | 0
  Conjuctival Staining | 0 | 0
  Bulbar Hyperemia | 0 | 0
  Limbal Hyperemia | 0 | 0
  Palpebral Hyperemia | 0 | 0
  Palpebral Roughness | 0 | 0
  Vascularization | 0 | 0
  "Other" Findings | 0 | 0

11. Secondary Outcome: Incidence of Adverse Events
Description: Cumulative incidence of adverse events.
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | Dual Focus Soft Contact Lens | Single Vision Soft Contact Lens
Number analyzed (Participants) | 58 | 60
participants
  Non-significant infiltrative event- device related | 0 | 2
  Blepharitis - not device related | 2 | 0
  Localized allergic reaction - device related | 0 | 1
  Localized allergic reaction-not device related | 0 | 1
  Non-significant-Other-Device related | 2 | 0
  Non-significant-Other- Not device related | 3 | 0
  Foreign Body -Device related | 1 | 0
  Corneal event -Device related | 3 | 0
  Corneal event- Not device related | 1 | 0
  Meibomianitis - Not device related | 2 | 0
  Significant adverse events | 0 | 0

12. Secondary Outcome: Incidence of Adverse Events
Description: Cumulative incidence of adverse events.
Time Frame: 24 months
Measure: Number; unit: participants
Arm/Group | Dual Focus Soft Contact Lens | Single Vision Soft Contact Lens
Number analyzed (Participants) | 55 | 60
participants
  Conjuctivitis - Not device related | 2 | 0
  Non-significant Other - Device related | 1 | 0
  Non-significant Other - Not device related | 0 | 3
  Non-significant infiltrative event Device related | 0 | 1
  Significant Adverse Events | 0 | 0

13. Secondary Outcome: Incidence of Adverse Events
Description: Cumulative incidence of adverse events.
Time Frame: 36 months
Measure: Number; unit: participants
Arm/Group | Dual Focus Soft Contact Lens | Single Vision Soft Contact Lens
Number analyzed (Participants) | 52 | 56
participants
  Conjuctivitis - Not device related | 0 | 1
  Non-significant Other - Device related | 0 | 1
  Non-significant Other - Not device related | 0 | 1
  Non-significant infiltrative event-no device relat | 1 | 0
  Corneal event- device related | 0 | 1
  Significant Adverse Events | 0 | 0

ADVERSE EVENTS:
Time Frame: From dispense of soft contact lenses till 36 months follow-up visit.
Arm/Group | Dual Focus Soft Contact Lens | Single Vision Soft Contact Lens
All-Cause Mortality (participants affected / at risk) | 0/70 | 0/74
Serious Adverse Events (participants affected / at risk) | 0/70 | 0/74
Other Adverse Events (participants affected / at risk) | 0/70 | 0/74

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2012-07-26): https://cdn.clinicaltrials.gov/large-docs/08/NCT01729208/Prot_000.pdf
  • Statistical Analysis Plan (2018-04-30): https://cdn.clinicaltrials.gov/large-docs/08/NCT01729208/SAP_001.pdf